CLINICAL TRIAL: NCT00763932
Title: A Multicenter, Open-Label Extension Study of the Long-Term Safety and Efficacy of Recombinant Human Acid α-Glucosidase (rhGAA) in Patients With Pompe Disease (Glycogen Storage Disease Type II) Who Were Previously Enrolled in Genzyme-Sponsored Enzyme Replacement Therapy Studies
Brief Title: Extension Study of Long-term Safety and Efficacy of Myozyme in Patients With Pompe Disease Who Were Previously Enrolled in Genzyme Sponsored Enzyme Replacement Therapy (ERT) Studies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLU02003
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Pompe Disease Infantile-Onset; Glycogen Storage Disease Type II
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Myozyme

INTERVENTIONS:
Biological: Myozyme — 10 mg/kg or 20 mg/kg qw OR 20 mg/kg or 40 mg/kg qow
  Other Names: Alglucosidase alfa

SUMMARY:
This extension study was to monitor the long-term safety and efficacy of rhGAA treatment in patients with infantile-onset Pompe disease who were previously treated with rhGAA derived from the Synpac cell line

ELIGIBILITY:
Inclusion Criteria:

* The patient was enrolled in Protocol AGLU-008-01, AGLU-009-02, or AGLU01502
* The patient's legal guardian(s) provided written informed consent prior to any study related procedures being performed
* The patient and his/her guardian(s) were able to comply with the clinical protocol, which required extensive clinical evaluations for an extended period of time.

Exclusion Criteria:

* Patients were excluded from this study if they did not meet the specific inclusion criteria, or if the patient experienced any unmanageable AE in Protocol AGLU-008-01, AGLU-009-02, or AGLU01502 (as determined and agreed upon by the Principal Investigator and Genzyme Corporation), due to Synpac rhGAA therapy, that would preclude continuing therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-04; Primary Completion 2006-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
The objective of this extension study was to monitor the long-term safety and efficacy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (8):
- United States (5):
  - Children's Hospital of Oakland, Oakland, California
  - Children's Hospital of Orange Country, Orange, California
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Institute for Genetic Medicine, Saint Peter's University Hospital, New Brunswick, New Jersey
  - New York University [NYU] School of Medicine, New York, New York
- France (2):
  - Pediatrique Hospital Debrousse, Lyon
  - Hôpital Porte Madeleine, Orléans
- The Morningside Clinic, Johannesburg, South Africa